CLINICAL TRIAL: NCT03745495
Title: Study to Determine the Effect of HIV Self-testing on the Uptake of and Retention in Pre-exposure Prophylaxis Service Among Older Adolescent Men Who Have Sex With Men and Transgender Women
Brief Title: HIV Self-Testing AND Uptake and Retention of PrEP Among Older Adolescent MSM and TGW
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: STANDUP-TEEN
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Men or Transgender Women Who Have Sex With Men
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 300 To determine the effect of HIVST on PrEP uptake among older adolescent MSM and TGW
- Group 2: 300 To determine the effect of HIVST on retention of older adolescent MSM and TGW in HIV service

SUMMARY:
This will be a prospective study that will enroll up to 600 older adolescent MSM and TGW from community-based clinics in Bangkok, Chonburi, Chiang Mai, and Songkhla.

DETAILED DESCRIPTION:
All eligible participants will be followed up at month 3, 6, 9, and 12; month 6 and 12 will be mandatory clinic visits, while month 3 and 9 will be either clinic or a virtual visits. For participants accepting PrEP, additional follow-up visit at month 1, 2, 4, and 5 will be appointed; all visits will be either clinic or virtual visits.

Study Sites

The study will take place at the following community-based clinics:

1. SWING DIC, Bangkok, Thailand
2. RSAT DIC, Bangkok, Thailand
3. SWING DIC, Chonburi, Thailand
4. Sister DIC, Chonburi, Thailand
5. Caremat DIC, Chiang Mai, Thailand
6. MPlus DIC, Chiang Mai, Thailand
7. RSAT DIC, Songkhla, Thailand

ELIGIBILITY:
Inclusion Criteria:

1. Thai nationality
2. Age 15-19 years old
3. Men or transgender women who have sex with men
4. HIV-negative at the time of screening
5. Have at least one of the following risks for HIV acquisition in the past 6 months:

   1. Any unprotected receptive anal sex with a male partner
   2. More than 5 male partners, regardless of condom use and serostatus
   3. Has had a bacterial sexually transmitted infection (STI)
   4. Any injected drug use
6. Calculated creatinine clearance (CrCl) ≥ 75 mL/min, as estimated by the Cockcroft- Gault equation
7. Alanine aminotransferase (ALT) ≤ 2.5 x ULN
8. Have signed the informed consent form

Exclusion Criteria:

1. HIV-positive
2. Hepatitis B infection as indicated by positive hepatitis B surface antigen (HBsAg) test at time of screening
3. Known allergy/sensitivity to tenofovir or emtricitabine

Ages: 15 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Approximately 600 older adolescent MSM and TGW
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Proportion of participants starting PrEP among those who use and do not use HIVST | 3 years
Proportion of participants taking PrEP retaining in care among those who use and do not use HIVST | 3 years

CONTACTS AND LOCATIONS:
Locations (7):
- Thailand (7):
  - 1.Swing Dic,, Bangkok
  - 2. Rsat Dic,, Bangkok
  - 5. Caremat DIC,, Chiang Mai
  - 6. MPlus DIC,, Chiang Mai
  - 3. Swing Dic,, Chon Buri
  - 4. Sister DIC,, Chon Buri
  - 7. Rsat Dic,, Songkhla